CLINICAL TRIAL: NCT06164223
Title: The Effect of the "VR Baby-Pump" Application Applied to Mothers Who Gave Birth Preterm on Their Breast Milk Expression Experience, Transition Process, and Milk Quantity: Randomized Controlled Study
Brief Title: Breast Milk Expression With Virtual Reality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Meltem Ozkaya, Research asistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Akdenizuniversityy
Record Dates: First submitted 2023-10-03; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Virtual Reality; Breast Milk Expression
Keywords: Transition to motherhood; Preterm birth; Breast milk expression experience; VR Baby Pump
MeSH Terms: conditions — Breast Milk Expression; Premature Birth

STUDY DESIGN:
Intervention Model Description: There are two Groups with parallel properties. The first group is the experimental group using virtual reality glasses.
  The second group is the control group without intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Group to which VR Baby Pump will be applied
  Interventions: Device: VR Baby Pump
- Control (No Intervention): An intervention will not be applied.

INTERVENTIONS:
Device: VR Baby Pump — VRBaby-Pump application is a video application specially prepared with virtual reality glasses and a milking pump placed inside a toy doll. In the video content, the mother is breastfeeding her baby on an armchair in the baby room prepared for a newborn baby.
  Arms: Experimental

SUMMARY:
The study is a randomized controlled study planned to determine the effect of the VRBaby-Pump application applied to mothers who gave birth preterm, on the mother's breast milk expression experience, transition process, and milk amount. In the study, the effectiveness of the VRBaby-Pump application will be evaluated based on evidence using the Breastfeeding Experience and Transition to Motherhood Scale. Stratified and block randomization methods will be used in the study. The study data will be collected from mothers who gave birth preterm at the Perinatology clinic of Health Sciences University (SBU) Antalya Training and Research Hospital between September and December 2023.

DETAILED DESCRIPTION:
Preterm labor is defined as births that occur before the 37th week of pregnancy is completed. While every 15 million babies worldwide are born prematurely, it is stated that 15 out of every 100 babies are premature in our country. Breast milk is the best source of nutrition for all newborn babies to complete their growth and development, and it is recommended that they be fed only with breast milk for the first six months; On the other hand, the rate of premature babies being exclusively breastfed for the first six months is quite low. It is perceived as an obligatory duty for mothers to not have their baby with them after birth, and to see a milking machine at their breast instead of their baby. Therefore, the transition to motherhood, the experiences they experience after birth, and the amount of milk the baby receives are affected. Nurses should support the mother who has given birth preterm to start and continue the lactation process, ensuring that the baby is fed with breast milk and has a positive experience with the transition to healthy motherhood. With the introduction of virtual reality applications into our lives in recent years, there are many areas of use in the field of health. Since it is not possible for mothers who give birth preterm to move from the hospital to the home environment with their babies immediately after birth, it is thought that by preparing a virtual baby and baby room, mothers will have good experiences during the lactation process and a healthy transition to motherhood, which will also lead to an increase in the amount of milk.

The study is a randomized controlled study planned to determine the effect of the VRBaby-Pump application applied to mothers who gave birth preterm, on the mother's milking experience, transition process, and milk amount. In the study, the effectiveness of the VRBaby-Pump application will be evaluated based on evidence using the Breastfeeding Experience and Transition to Motherhood Scale. Stratified and block randomization methods will be used in the study. The study data will be collected from mothers who gave birth preterm at the Perinatology Clinic of Health Sciences University (SBU) Antalya Training and Research Hospital between September and December 2023. This study will be the first nursing study on this subject in both national and international literature. As a result of this study, the milking experience of mothers who gave birth preterm, the transition to motherhood, and the amount of milk will be determined, and a new milk-selling virtual reality program will be offered to mothers who give birth preterm.

ELIGIBILITY:
Inclusion Criteria:

1. Having given birth before the 37th week of pregnancy
2. The baby is in the neonatal intensive care unit
3. Being on postpartum day 0
4. Being milked
5. Being a citizen of the Republic of Türkiye,

Exclusion Criteria:

1. Loss of the newborn
2. Leaving the newborn from the intensive care unit before the second postpartum day
3. The mother has a condition that prevents breastfeeding
4. The mother states that she feels discomfort (nausea, disorientation, etc.) when the application begins.
5. Those with vision and hearing problems
6. Those with a psychiatric diagnosis
7. Those who are not capable of using virtual reality glasses
8. Those who watched the video while only one breast was being pumped (those who watched only 15 minutes)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 88 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the transition process to motherhood of mothers who gave birth preterm | Postpartum 2nd day
  transition to positive motherhood, It will use the Transition of Motherhood Scale to do an evaluation
Evaluation of the breast milk expression experience of mothers who gave birth preterm | Postpartum 2nd day
  positive breast milk expression experience, It will use the Breast Milk Expression Experience Scale to do an evaluation
Evaluation of milk quantity of mothers who gave birth preterm | Postpartum 2nd day
  high amount of breast milk, It will use the Daily Breast Milk Form to do an evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Oznur Korukcu, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No